CLINICAL TRIAL: NCT00966810
Title: Allogeneic Stem Cell Transplantation in CML With Partial T Cell Depletion and Preemptive Donor Lymphocyte Infusion.
Brief Title: Allogeneic Stem Cell Transplantation in CML With Partial T Cell Depletion
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Tsila Zuckerman, MD, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML ASCTCTIL
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2009-08-27 (Estimated); Status verified 2009-01

CONDITIONS: Philadelphia Chromosome-positive Chronic Myelocytic Leukemia
Keywords: chronic myelocytic leukemia; allogeneic stem cell transplantation; T cell depletion; donor lymphocyte infusion; GvHD; transplant related mortality
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CML allogeneic stem cell transplantation (Experimental): Patients with chronic myeloid leukemia suitable for allogeneic stem cell transplantation with a matched related donor.
  Interventions: Procedure: Stem cell transplantation

INTERVENTIONS:
Procedure: Stem cell transplantation — Patients were conditioned with oral busulfan 12mg/kg (days -6 to -4), cyclophosphamide 120mg/kg (days -3,-2), rabbit antithymocytic globulin, (Fresenius, Bad Hamburg, Germany) 25mg/kg (days -5 to -1) and fludarabine 200 mg/kg (days -7 to-3). CD34 cells were positively selected using anti-CD34 antibody conjugated to iron-dextran microbeads using CliniMACS device (Miltenyi Biotech, Bergisch Gladbach, Germany) with an aim to collect > 5.0 x 106 CD34 cells/kg. DLI was administered in escalating dose regimen starting from 3 x 106 cells/kg followed as necessary by 1 x 107 cells/kg, 5 x 107 cells/kg and 1 x 108 cells/kg.
  Other Names: HSCT

SUMMARY:
Allogeneic stem cell transplantation, the only known curative modality for CML, was abandoned in recent years for a very effective and much less toxic targeted therapy with the tyrosine kinase inhibitors (TKIs). However, approximately one third of patients still need another treatment including stem cell transplantation. The study protocol comprised a cohort of consecutive patients with CML who received allogeneic stem cell transplantation using partial T cell depletion, with no post-transplant GvHD prophylaxis. Forty consecutive patients with CML underwent allogeneic stem cell transplantation from a matched sibling using partial T cell depletion (TCD), in a single institution. Escalated dose of donor lymphocyte infusion (DLI) was given in case of either relapse or presence of minimal residual disease (MRD) as detected by cytogenetic or molecular analysis.

The purpose of the study is to decrease transplant-related toxicity.

DETAILED DESCRIPTION:
Patients were conditioned with oral busulfan 12mg/kg (days -6 to -4), cyclophosphamide 120mg/kg (days -3,-2), rabbit antithymocytic globulin, (Fresenius, Bad Hamburg, Germany) 25mg/kg (days -5 to -1) and fludarabine 200 mg/kg (days -7 to-3). Final busulfan dose was individually determined based on measurements of serum busulfan levels with a target dose of 850-1400 microM x minute.

Transplants were performed in reverse isolation rooms equipped with high-efficiency particulate air filtration systems (HEPA). No post-transplant GvHD prophylaxis was given. Post-transplant infection prophylaxis consisted of acyclovir, itraconazole, trimethoprim-sulfamethoxazole and penicillin VK. Cytomegalovirus (CMV) status was determined weekly using PCR for CMV-DNA and pp65 antigenemia in blood leukocytes, followed by preemptive ganciclovir administration when positive.

Donors Donors were human leukocyte antigen (HLA) A,B,C serologically matched and DR and DQ molecularly matched siblings. Donor stem cells were collected following mobilization with 10 µg/kg/day G-CSF, given subcutaneously for 5 consecutive days. CD34 cells were positively selected using anti-CD34 antibody conjugated to iron-dextran microbeads using CliniMACS device (Miltenyi Biotech, Bergisch Gladbach, Germany) with an aim to collect > 5.0 x 106 CD34 cells/kg.

Disease monitoring Following transplant, all patients were under close surveillance for the presence of minimal residual disease (MRD) using cytogenetic analysis and PCR for the detection of BCR/ABL transcripts. Bone marrow and peripheral blood samples were examined every 3 months in the first year post transplant and every 3-6 months in the subsequent years.

PCR method: RQ-PCR was performed according to the Europe Against Cancer (EAC) protocol.19 The BCR-ABL and ABL copy numbers were calculated by comparing with the standard curve generated using IPSOGEN FusionQuant Standards. The results of quantifying BCR-ABL transcripts were expressed as percentage ratios relative to total ABL transcripts.

A minimum number of 1x104 copies of ABL is the lower limit below which a negative RT-PCR was considered unreliable. In the molecular biology laboratory of the Rambam Health Care Campus the sensitivity for quantitative Q-PCR is (10-5).

Donor leukocyte infusion (DLI). DLI was administered in escalating dose regimen starting from 3 x 106 cells/kg followed as necessary by 1 x 107 cells/kg, 5 x 107 cells/kg and 1 x 108 cells/kg.

DLI was used in case of persistence/reappearance of BCR-ABL transcripts starting from 6 months post transplant onward. In instances where more than 1 DLI was administered the successive escalated dose was given at ≥ 3-month intervals as dictated by MRD follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic phase CML by hematological, cytogenetic and molecular studies.
* Age >18
* Candidates for allogeneic stem cell transplantation
* Available matched related donor

Exclusion Criteria:

* Age< 18 years
* Other malignancy
* Decreased cardiac function (by echo), reduced pulmonary function (decreased DLCO, FEV1), abnormal kidney function (creatinine > 1.5 N), abnormal liver function (AST, ALT >2N)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1999-12; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | The outcome is assessed at the end of transplant and every 3-6 months thereafter continuously.

SECONDARY OUTCOMES:
Overall survival | Every 3-6 months after transplant continuously.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M Rowe, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

REFERENCES:
- [Background] O'Brien SG, Guilhot F, Larson RA, Gathmann I, Baccarani M, Cervantes F, Cornelissen JJ, Fischer T, Hochhaus A, Hughes T, Lechner K, Nielsen JL, Rousselot P, Reiffers J, Saglio G, Shepherd J, Simonsson B, Gratwohl A, Goldman JM, Kantarjian H, Taylor K, Verhoef G, Bolton AE, Capdeville R, Druker BJ; IRIS Investigators. Imatinib compared with interferon and low-dose cytarabine for newly diagnosed chronic-phase chronic myeloid leukemia. N Engl J Med. 2003 Mar 13;348(11):994-1004. doi: 10.1056/NEJMoa022457. PMID 12637609
- [Background] Hughes TP, Kaeda J, Branford S, Rudzki Z, Hochhaus A, Hensley ML, Gathmann I, Bolton AE, van Hoomissen IC, Goldman JM, Radich JP; International Randomised Study of Interferon versus STI571 (IRIS) Study Group. Frequency of major molecular responses to imatinib or interferon alfa plus cytarabine in newly diagnosed chronic myeloid leukemia. N Engl J Med. 2003 Oct 9;349(15):1423-32. doi: 10.1056/NEJMoa030513. PMID 14534335
- [Background] Druker BJ, Guilhot F, O'Brien SG, Gathmann I, Kantarjian H, Gattermann N, Deininger MW, Silver RT, Goldman JM, Stone RM, Cervantes F, Hochhaus A, Powell BL, Gabrilove JL, Rousselot P, Reiffers J, Cornelissen JJ, Hughes T, Agis H, Fischer T, Verhoef G, Shepherd J, Saglio G, Gratwohl A, Nielsen JL, Radich JP, Simonsson B, Taylor K, Baccarani M, So C, Letvak L, Larson RA; IRIS Investigators. Five-year follow-up of patients receiving imatinib for chronic myeloid leukemia. N Engl J Med. 2006 Dec 7;355(23):2408-17. doi: 10.1056/NEJMoa062867. PMID 17151364
- [Background] Jabbour E, Cortes JE, Kantarjian HM. Molecular monitoring in chronic myeloid leukemia: response to tyrosine kinase inhibitors and prognostic implications. Cancer. 2008 May 15;112(10):2112-8. doi: 10.1002/cncr.23427. PMID 18348294
- [Background] de Lavallade H, Apperley JF, Khorashad JS, Milojkovic D, Reid AG, Bua M, Szydlo R, Olavarria E, Kaeda J, Goldman JM, Marin D. Imatinib for newly diagnosed patients with chronic myeloid leukemia: incidence of sustained responses in an intention-to-treat analysis. J Clin Oncol. 2008 Jul 10;26(20):3358-63. doi: 10.1200/JCO.2007.15.8154. Epub 2008 Jun 2. PMID 18519952
- [Background] Gratwohl A, Hermans J, Goldman JM, Arcese W, Carreras E, Devergie A, Frassoni F, Gahrton G, Kolb HJ, Niederwieser D, Ruutu T, Vernant JP, de Witte T, Apperley J. Risk assessment for patients with chronic myeloid leukaemia before allogeneic blood or marrow transplantation. Chronic Leukemia Working Party of the European Group for Blood and Marrow Transplantation. Lancet. 1998 Oct 3;352(9134):1087-92. doi: 10.1016/s0140-6736(98)03030-x. PMID 9798583
- [Background] Passweg JR, Walker I, Sobocinski KA, Klein JP, Horowitz MM, Giralt SA; Chronic Leukemia Study Writing Committee of the International Bone Marrow Transplant Registry. Validation and extension of the EBMT Risk Score for patients with chronic myeloid leukaemia (CML) receiving allogeneic haematopoietic stem cell transplants. Br J Haematol. 2004 Jun;125(5):613-20. doi: 10.1111/j.1365-2141.2004.04955.x. PMID 15147377
- [Background] Baccarani M, Saglio G, Goldman J, Hochhaus A, Simonsson B, Appelbaum F, Apperley J, Cervantes F, Cortes J, Deininger M, Gratwohl A, Guilhot F, Horowitz M, Hughes T, Kantarjian H, Larson R, Niederwieser D, Silver R, Hehlmann R; European LeukemiaNet. Evolving concepts in the management of chronic myeloid leukemia: recommendations from an expert panel on behalf of the European LeukemiaNet. Blood. 2006 Sep 15;108(6):1809-20. doi: 10.1182/blood-2006-02-005686. Epub 2006 May 18. PMID 16709930
- [Background] Goldman JM. How I treat chronic myeloid leukemia in the imatinib era. Blood. 2007 Oct 15;110(8):2828-37. doi: 10.1182/blood-2007-04-038943. Epub 2007 Jul 12. PMID 17626839
- [Derived] Zuckerman T, Katz T, Haddad N, Fineman R, Dann EJ, Avivi I, Ofran Y, Gavish I, Faibish T, Sahar D, Hertz E, Sabo E, Reisner Y, Rowe JM. Allogeneic stem cell transplantation for patients with chronic myeloid leukemia: risk stratified approach with a long-term follow-up. Am J Hematol. 2012 Sep;87(9):875-9. doi: 10.1002/ajh.23263. Epub 2012 Jul 27. PMID 22847303